CLINICAL TRIAL: NCT05141214
Title: Virtual Reality as a Dietary Education Adjunct for Pediatric Patients With Obesity: A Pragmatic, Randomized Pilot Study
Brief Title: Virtual Reality as a Dietary Education Adjunct for Pediatric Patients With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 63298
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Diabetes
Keywords: Virtual Reality
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Consult with Virtual Reality (intervention) (Active Comparator): Those in the VR group will receive the same educational dietary review by the registered dietician, and additionally participate in a VR experience through an application called Chaos Café. In Chaos Café, patients are immersed into a computer-generated kitchen environment. A humorous robotic chef serves children different food groups. Gameplay is advanced by choosing healthy foods, while eating unhealthy foods does not advance the application.
  Interventions: Behavioral: Virtual Reality Application
- Dietary Consult without Virtual Reality (SOC) (No Intervention): Those in the SOC group will have the typical appointment, which includes a review of healthy diet choices with a registered dietitian and follow up according to clinic's SOC.

INTERVENTIONS:
Behavioral: Virtual Reality Application — In VR application, Chaos Café, patients are immersed into a computer-generated kitchen environment. A humorous robotic chef serves children different food groups. Gameplay is advanced by choosing healthy foods, while eating unhealthy foods does not advance the application.
  Arms: Dietary Consult with Virtual Reality (intervention)

SUMMARY:
Childhood obesity is a national crisis, effecting up to 1 in 5 of children in the US. In the Lucile Packard Children's Hospital Pediatric Weight Management Clinic, the investigators educate parents and caregivers about the importance of dietary modification. In addition to physician guidance, the investigators partner with registered dieticians to counsel families during an hour-long interview. However, traditional methods of education are limited by long-term recall. A typical person only recalls 2- 3% of didactic content after a period of 30 days. In order to improve recall and increase involvement of our pediatric patients in their own dietary modifications, the investigators propose a pragmatic, randomized pilot study investigating the effectiveness of Virtual Reality (VR) in changing dietary choices and improving recall.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-18 years of age
* Able to consent or have parental consent
* Diagnosis of Obesity Grade 1, 2 and 3 at LPCH/SHC facilities

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Visual Problems

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Immediate behavior modification | Duration of appointment, typically 2-3 hours
  Immediate behavior modification will be assessed by comparing the selection of an appointment exit reward the end of the study visit. Participants will be presented with two options, either a bag of chips or a healthier alternative. Selection of reward will be recorded.

SECONDARY OUTCOMES:
Pediatric Adapted Liking Survey | Duration of appointment, typically 2-3 hours
  The survey uses a continuous scale from -100 to 100 to indicate patients' like or dislike of certain foods. The survey was completed by participants after their dietary counseling. The responses were categorized into seven groups, 3 negative, 1 neutral, and 3 positive. -3=[-100,-67], -2=[-66,-34], -1=[-33,-1], 0=0, 1=[1,33], 2=[34,66], 3=[67,100]. Likability of foods were also categorized into fruits, fatty/salty/sugary (FSS), proteins and vegetables.
Nutritional knowledge survey | Duration of appointment, typically 2-3 hours
  15-item survey based on the counseling sessions with questions such as "If I have vegetables at home, a healthy way to eat them would be: a) fresh, b) fried, c)with cheese dip, d)in a smoothie"
Satisfaction Survey | Duration of appointment, typically 2-3 hours
  5-point satisfaction survey for participants who completed VR experience with questions such as "The technology helps me remember what good food choices are (select one option): (1) Not at all, (2), (3) A little bit, (4), (5) A lot"

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No